CLINICAL TRIAL: NCT03699553
Title: Positive Affect Regulation as Adjuvant to Integrative Therapies for Chronic Pain: Development of the LARKSPUR Clinic-Based Intervention
Brief Title: Lessons in Affect Regulation to Keep Stress and Pain UndeR Control (LARKSPUR R34)
Acronym: LARKSPUR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: BraveNet (Other)
Responsible Party: Principal Investigator, Judith Moskowitz, Professor, Northwestern University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SP0042991
Record Dates: First submitted 2018-07-19; First posted 2018-10-09 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Chronic Pain; Musculoskeletal Pain
Keywords: online intervention; chronic pain; positive emotion; affective science
MeSH Terms: conditions — Chronic Pain; Musculoskeletal Pain

STUDY DESIGN:
Intervention Model Description: 40 participants will be randomized to the LARKSPUR Study. 20 will receive the online intervention and 20 will report their daily emotions for the same duration as the intervention. The 20 individuals assigned to the emotion reporting (control group) arm will receive the online intervention after completing the final assessment, 12 weeks after baseline.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will receive the online LARKSPUR intervention which lasts about 5-6 weeks, receiving the positive emotions skills through the website, and logging on to the website for about 5-10 minutes each day for that period. Assessments will be taken at baseline, post-intervention (8 weeks after the baseline), and 12 weeks after baseline (1 month post intervention).
  Interventions: Behavioral: LARKSPUR; Online Positive Emotions Skills for Individuals with Chronic Musculoskeletal Pain
- Emotion Reporting Control (Active Comparator): Participants will report their emotions for 5-6 weeks by logging on to the website for about 5 minutes each day. Assessments will be taken at baseline, 8 weeks after baseline, and 12 weeks after baseline. After 12 weeks, participants will receive access to the LARKSPUR intervention online.
  Interventions: Behavioral: Emotion Reporting Control Group

INTERVENTIONS:
Behavioral: LARKSPUR; Online Positive Emotions Skills for Individuals with Chronic Musculoskeletal Pain — 8 positive emotion skills taught over 5-6 weeks to help individuals cope with chronic pain and stress.
  Arms: Intervention
Behavioral: Emotion Reporting Control Group — Attention matched control condition, participants will report their daily emotions over 5-6 weeks online.
  Arms: Emotion Reporting Control

SUMMARY:
Chronic pain affects millions of Americans but integrative as well as conventional treatments fall short in terms of alleviating this pain. The investigators are testing a tailored online positive affect skills intervention through a high-quality, randomized controlled trial for people with chronic musculoskeletal pain. The proposed work holds promise as an effective, low cost, easily disseminated intervention to help people cope with chronic pain, decrease depression and distress that pose barriers to optimal adherence, and potentially boost the efficacy of integrative as well as conventional pain treatments.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and over
* Current patient at Northwestern Memorial Hospital
* Seeking treatment for chronic musculoskeletal pain at the Northwestern Osher Center for Integrative Medicine. Pain will be defined as persisting for at least the past three months with an average level over the past month of at least 4 of 10 on a numerical rating scale, including back pain, neck pain/cervicalgia, knee pain, other joint pain (hips, ankles), fibromyalgia, osteoarthritis and rheumatoid arthritis.
* Fluent in the English language
* Have a working email address
* Have reliable Internet access in order to access the website online

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Retention to the LARKSPUR Study from baseline to 8 weeks post baseline | 8 weeks; from baseline to 8 weeks post baseline
  Retention will be defined as responding to the assessments at baseline and at 8 weeks post baseline
Retention to the LARKSPUR Study from baseline to 12 weeks post baseline | 12 weeks; from baseline to 12 weeks post baseline
  Retention will be defined as responding to the assessments at baseline and at 12 weeks post baseline

SECONDARY OUTCOMES:
Self-Reported Medication use at baseline | Administered at baseline
  Measuring medication use by asking: "Have you used any prescription or non-prescription medication for your pain in the last 7 days?" with a Yes-No response. If "Yes" is selected, options include 13 types of medications as response options, with 2 follow-up question for each medication selected: "How many milligrams (mg) per pill, if you know it?" and "What is the average number of pills per day?"
Self-Reported Medication use at 8 weeks post baseline | Administered at 8 weeks post baseline
  Measuring medication use by asking: "Have you used any prescription or non-prescription medication for your pain in the last 7 days?" with a Yes-No response. If "Yes" is selected, options include 13 types of medications as response options, with 2 follow-up question for each medication selected: "How many milligrams (mg) per pill, if you know it?" and "What is the average number of pills per day?"
Self-Reported Medication use at 12 weeks post baseline | Administered at 12 weeks post baseline
  Measuring medication use by asking: "Have you used any prescription or non-prescription medication for your pain in the last 7 days?" with a Yes-No response. If "Yes" is selected, options include 13 types of medications as response options, with 2 follow-up question for each medication selected: "How many milligrams (mg) per pill, if you know it?" and "What is the average number of pills per day?"
Modified Differential Emotions Scale (mDES) | Administered daily for 5 weeks of the intervention period
  Measuring positive and negative affect through a 26-item modified version of the Differential Emotions Scale with the anchor: "How much have you felt each of these emotions over the PAST DAY?" with items including "amused or fun-loving" "angry, irritated, or frustrated" and "anxious or scared." Response scale is from 1 Not at all to 9 All the time.
Daily Inventory of Stressful Events (DISE) | Administered daily for 5 weeks of the intervention period
  Measuring stress through a 7-item scale with the following anchor: "Over the PAST DAY, have you…" and the items include: "Had an argument or disagreement with someone?" and "Almost had an argument or disagreement but decided to let it pass to avoid disagreement?" The response scale is from 0 Didn't happen to 4 Very Stressful.
Pain Level, measured by a single-item pain question | Administered daily for 5 weeks of the intervention period
  Measuring daily pain level through the single-item: "What is your level of pain right now?" Response items range from 0 No Pain to 10 Pain as bad as you can imagine.
Positive Affect using the NIH Toolbox for Positive Affect, Short-Form (Baseline) | Administered at baseline
  A 16-item measure that asks: "In the past 7 days…" and there are 15 items such as "I felt cheerful" "I felt attentive" "I felt delighted" "I felt happy." The response scale ranges from 1 Not at all to 5 Very much.
Positive Affect using the NIH Toolbox for Positive Affect, Short-Form (8 weeks post baseline) | Administered at 8 weeks post baseline
  A 16-item measure that asks: "In the past 7 days…" and there are 15 items such as "I felt cheerful" "I felt attentive" "I felt delighted" "I felt happy." The response scale ranges from 1 Not at all to 5 Very much.
Positive Affect using the NIH Toolbox for Positive Affect, Short-Form (12 weeks post baseline) | Administered at 12 weeks post baseline
  A 16-item measure that asks: "In the past 7 days…" and there are 15 items such as "I felt cheerful" "I felt attentive" "I felt delighted" "I felt happy." The response scale ranges from 1 Not at all to 5 Very much.
Emotional Support at baseline using the NIH Toolbox for Emotional Support | Administered at baseline
  Measuring emotional support through the 4-item NIH Toolbox measure for emotional support (4a) with questions such as "I have someone who will listen to me when I need to talk" and "I have someone to confide in or talk about myself or my problems." The response is on a 5-point scale from Never to Always.
Emotional Support at 8 weeks post baseline using the NIH Toolbox for Emotional Support | Administered at 8 weeks post baseline
  Measuring emotional support through the 4-item NIH Toolbox measure for emotional support (4a) with questions such as "I have someone who will listen to me when I need to talk" and "I have someone to confide in or talk about myself or my problems." The response is on a 5-point scale from Never to Always.
Emotional Support at 12 weeks post baseline using the NIH Toolbox for Emotional Support | Administered at 12 weeks post baseline
  Measuring emotional support through the 4-item NIH Toolbox measure for emotional support (4a) with questions such as "I have someone who will listen to me when I need to talk" and "I have someone to confide in or talk about myself or my problems." The response is on a 5-point scale from Never to Always.
Physical Function at Baseline through the PROMIS measure for physical function | Administered at baseline
  Measuring physical function through the 4-item PROMIS Short-From v2.0 - Physical Function 4a. Questions include: "Are you able to do chores such as vacuuming or yard work?" or "Are you able to go up and down stairs at a normal pace?" Responses are on a 5-point scale from "Without any difficulty" to "Unable to do."
Physical Function at 8 weeks post baseline through the PROMIS measure for physical function | Administered at 8 weeks post baseline
  Measuring physical function through the 4-item PROMIS Short-From v2.0 - Physical Function 4a. Questions include: "Are you able to do chores such as vacuuming or yard work?" or "Are you able to go up and down stairs at a normal pace?" Responses are on a 5-point scale from "Without any difficulty" to "Unable to do."
Physical Function at 12 weeks post baseline through the PROMIS measure for physical function | Administered at 12 weeks post baseline
  Measuring physical function through the 4-item PROMIS Short-From v2.0 - Physical Function 4a. Questions include: "Are you able to do chores such as vacuuming or yard work?" or "Are you able to go up and down stairs at a normal pace?" Responses are on a 5-point scale from "Without any difficulty" to "Unable to do."
Pain on average over 7 days at baseline through a single-item question | Administered at baseline
  Measuring pain on average over the past 7 days with a single-item question: "In the past 7 days, how would you rate your pain on average?" The response scale ranges from 0 No pain to 10 Pain as bad as you can imagine.
Pain on average over 7 days at 8 weeks post baseline through a single-item question | Administered at 8 weeks post baseline
  Measuring pain on average over the past 7 days with a single-item question: "In the past 7 days, how would you rate your pain on average?" The response scale ranges from 0 No pain to 10 Pain as bad as you can imagine.
Pain on average over 7 days at 12 weeks post baseline through a single-item question | Administered at 12 weeks post baseline
  Measuring pain on average over the past 7 days with a single-item question: "In the past 7 days, how would you rate your pain on average?" The response scale ranges from 0 No pain to 10 Pain as bad as you can imagine.
Depression at baseline using the PROMIS measure | Administered at baseline
  Measuring depression using the PROMIS Short-Form v1.0-Depression 4a with 4 items including: "In the past 7 days I felt worthless" and "In the past 7 days I felt helpless." The 5-point response scale ranges from Never to Always.
Depression at 8 weeks post baseline using the PROMIS measure | Administered at 8 weeks post baseline
  Measuring depression using the PROMIS Short-Form v1.0-Depression 4a with 4 items including: "In the past 7 days I felt worthless" and "In the past 7 days I felt helpless." The 5-point response scale ranges from Never to Always.
Depression at 12 weeks post baseline using the PROMIS measure | Administered at 12 weeks post baseline
  Measuring depression using the PROMIS Short-Form v1.0-Depression 4a with 4 items including: "In the past 7 days I felt worthless" and "In the past 7 days I felt helpless." The 5-point response scale ranges from Never to Always.
Anxiety at baseline using the PROMIS measure | Administered at baseline
  Measuring anxiety using the PROMIS Short-Form v1.0-Anxiety 4a with 4 items such as "In the past 7 days I felt fearful" and "In the past 7 days I found it hard to focus on anything other than my anxiety." The 5-point response scale ranges from Never to Always.
Anxiety at 8 weeks post baseline using the PROMIS measure | Administered at 8 weeks post baseline
  Measuring anxiety using the PROMIS Short-Form v1.0-Anxiety 4a with 4 items such as "In the past 7 days I felt fearful" and "In the past 7 days I found it hard to focus on anything other than my anxiety." The 5-point response scale ranges from Never to Always.
Anxiety at 12 weeks post baseline using the PROMIS measure | Administered at 12 weeks post baseline
  Measuring anxiety using the PROMIS Short-Form v1.0-Anxiety 4a with 4 items such as "In the past 7 days I felt fearful" and "In the past 7 days I found it hard to focus on anything other than my anxiety." The 5-point response scale ranges from Never to Always.
Pain Intensity at baseline using the PROMIS measure | Administered at baseline
  Measuring pain intensity using the PROMIS Scale v.1.0- Pain Intensity 3a which consists of 3 questions with the anchor: "In the past 7 days…" and the items include "How intense was your pain at its worst?" "How intense was your average pain?" and "What is your level of pain right now?" The 5-item response scale ranges from "Had no pain" to "Very severe."
Pain Intensity at 8 weeks post baseline using the PROMIS measure | Administered at 8 weeks post baseline
  Measuring pain intensity using the PROMIS Scale v.1.0- Pain Intensity 3a which consists of 3 questions with the anchor: "In the past 7 days…" and the items include "How intense was your pain at its worst?" "How intense was your average pain?" and "What is your level of pain right now?" The 5-item response scale ranges from "Had no pain" to "Very severe."
Pain Intensity at 12 weeks post baseline using the PROMIS measure | Administered at 12 weeks post baseline
  Measuring pain intensity using the PROMIS Scale v.1.0- Pain Intensity 3a which consists of 3 questions with the anchor: "In the past 7 days…" and the items include "How intense was your pain at its worst?" "How intense was your average pain?" and "What is your level of pain right now?" The 5-item response scale ranges from "Had no pain" to "Very severe."
Pain interference at baseline using the PROMIS measure | Administered at baseline
  Measuring pain interference using the PROMIS SF v1.0 - pain Interference 8a with the anchor: "In the past 7 days…" with 8 items including: "How much did pain interfere with your day to day activities?" "How much did pain interfere with work around the home?" or "How much did pain interfere with your ability to participate in social activities?" The 5-item response scale ranges from "Not at all" to "Very much."
Pain interference at 8 weeks post baseline using the PROMIS measure | Administered at 8 weeks post baseline
  Measuring pain interference using the PROMIS SF v1.0 - pain Interference 8a with the anchor: "In the past 7 days…" with 8 items including: "How much did pain interfere with your day to day activities?" "How much did pain interfere with work around the home?" or "How much did pain interfere with your ability to participate in social activities?" The 5-item response scale ranges from "Not at all" to "Very much."
Pain interference at 12 weeks post baseline using the PROMIS measure | Administered at 12 weeks post baseline
  Measuring pain interference using the PROMIS SF v1.0 - pain Interference 8a with the anchor: "In the past 7 days…" with 8 items including: "How much did pain interfere with your day to day activities?" "How much did pain interfere with work around the home?" or "How much did pain interfere with your ability to participate in social activities?" The 5-item response scale ranges from "Not at all" to "Very much."
Pain Self Efficacy at baseline (PSEQ) | Administered at baseline
  Measuring pain self efficacy using the Pain Self Efficacy Questionnaire (PSEQ) which has 10 items with the anchor: "Please rate how confident you are that you can do the following things at present, despite the pain." Items include: "I can enjoy things, despite the pain." "I can cope with my pain in most situations." "I can cope with my pain without medication." The response scale ranges from 0 Not at all Confident to 6 Completely Confident.
Pain Self Efficacy at 8 weeks post baseline (PSEQ) | Administered at 8 weeks post baseline
  Measuring pain self efficacy using the Pain Self Efficacy Questionnaire (PSEQ) which has 10 items with the anchor: "Please rate how confident you are that you can do the following things at present, despite the pain." Items include: "I can enjoy things, despite the pain." "I can cope with my pain in most situations." "I can cope with my pain without medication." The response scale ranges from 0 Not at all Confident to 6 Completely Confident.
Pain Self Efficacy at 12 weeks post baseline (PSEQ) | Administered at 12 weeks post baseline
  Measuring pain self efficacy using the Pain Self Efficacy Questionnaire (PSEQ) which has 10 items with the anchor: "Please rate how confident you are that you can do the following things at present, despite the pain." Items include: "I can enjoy things, despite the pain." "I can cope with my pain in most situations." "I can cope with my pain without medication." The response scale ranges from 0 Not at all Confident to 6 Completely Confident.
Pain resilience at baseline | Administered at baseline
  Measuring pain resilience using the 14 item Pain Resilience Scale. The anchor is: "When faced with intense or prolonged pain…" Items include "I get back out there" "I push through it" "I keep a positive attitude" and "I try to stay relaxed." The 5-item response scale ranges from "0 Not at all" to "4 All the time."
Pain resilience at 8 weeks post baseline | Administered at 8 weeks post baseline
  Measuring pain resilience using the 14 item Pain Resilience Scale. The anchor is: "When faced with intense or prolonged pain…" Items include "I get back out there" "I push through it" "I keep a positive attitude" and "I try to stay relaxed." The 5-item response scale ranges from "0 Not at all" to "4 All the time."
Pain resilience at 12 weeks post baseline | Administered at 12 weeks post baseline
  Measuring pain resilience using the 14 item Pain Resilience Scale. The anchor is: "When faced with intense or prolonged pain…" Items include "I get back out there" "I push through it" "I keep a positive attitude" and "I try to stay relaxed." The 5-item response scale ranges from "0 Not at all" to "4 All the time."
Pain catastrophizing at baseline | Administered at baseline
  Measuring pain catastrophizing using the Pain Catastrophizing Scale which has 13 items with the anchor: "When I'm in pain…" Items include: "I feel I can't go on." "I feel I can't stand it anymore." "I keep thinking about how much it hurts." The response scale ranges from 0 Not al all to 4 All the Time.
Pain catastrophizing at 8 weeks post baseline | Administered at 8 weeks post baseline
  Measuring pain catastrophizing using the Pain Catastrophizing Scale which has 13 items with the anchor: "When I'm in pain…" Items include: "I feel I can't go on." "I feel I can't stand it anymore." "I keep thinking about how much it hurts." The response scale ranges from 0 Not al all to 4 All the Time.
Pain catastrophizing at 12 weeks post baseline | Administered at 12 weeks post baseline
  Measuring pain catastrophizing using the Pain Catastrophizing Scale which has 13 items with the anchor: "When I'm in pain…" Items include: "I feel I can't go on." "I feel I can't stand it anymore." "I keep thinking about how much it hurts." The response scale ranges from 0 Not al all to 4 All the Time.
Patient adherence at baseline | Administered at baseline
  Measuring patient adherence to medical recommendations using the Medical Outcomes Study (MOS) Measures of Patient Adherence. The instrument has 5 items. The first four items ask questions like "I had a hard time doing what the doctor suggested I do… " or "I was unable to do what was necessary to follow my doctor's treatment plans…." The 5th item asks: "Generally speaking, how often during the past 4 weeks were you able to do what the doctor told you?" The 6-item response scale ranges from None of the time to All of the time.
Patient adherence at 8 weeks post baseline | Administered at 8 weeks post baseline
  Measuring patient adherence to medical recommendations using the Medical Outcomes Study (MOS) Measures of Patient Adherence. The instrument has 5 items. The first four items ask questions like "I had a hard time doing what the doctor suggested I do… " or "I was unable to do what was necessary to follow my doctor's treatment plans…." The 5th item asks: "Generally speaking, how often during the past 4 weeks were you able to do what the doctor told you?" The 6-item response scale ranges from None of the time to All of the time.
Patient adherence at 12 weeks post baseline | Administered at 12 weeks post baseline
  Measuring patient adherence to medical recommendations using the Medical Outcomes Study (MOS) Measures of Patient Adherence. The instrument has 5 items. The first four items ask questions like "I had a hard time doing what the doctor suggested I do… " or "I was unable to do what was necessary to follow my doctor's treatment plans…." The 5th item asks: "Generally speaking, how often during the past 4 weeks were you able to do what the doctor told you?" The 6-item response scale ranges from None of the time to All of the time.
Sleep disturbance at baseline using the PROMIS measure | Administered at baseline
  Measuring sleep disturbance using the 4-item PROMIS Short Form v.1.0 - Sleep Disturbance 4a with the anchor: "In the past 7 days…" Three of the items are: "My sleep was refreshing" "I had a problem with my sleep" and "I had difficulty falling asleep." The 5-item response scale ranges from "Not at all" to "Very much." The fourth question is: "My sleep quality was…" with the 5-item response scale ranging from "Very poor" to "Very good."
Sleep disturbance at 8 weeks post baseline using the PROMIS measure | Administered at 8 weeks post baseline
  Measuring sleep disturbance using the 4-item PROMIS Short Form v.1.0 - Sleep Disturbance 4a with the anchor: "In the past 7 days…" Three of the items are: "My sleep was refreshing" "I had a problem with my sleep" and "I had difficulty falling asleep." The 5-item response scale ranges from "Not at all" to "Very much." The fourth question is: "My sleep quality was…" with the 5-item response scale ranging from "Very poor" to "Very good."
Sleep disturbance at 12 weeks post baseline using the PROMIS measure | Administered at 12 weeks post baseline
  Measuring sleep disturbance using the 4-item PROMIS Short Form v.1.0 - Sleep Disturbance 4a with the anchor: "In the past 7 days…" Three of the items are: "My sleep was refreshing" "I had a problem with my sleep" and "I had difficulty falling asleep." The 5-item response scale ranges from "Not at all" to "Very much." The fourth question is: "My sleep quality was…" with the 5-item response scale ranging from "Very poor" to "Very good."

OTHER OUTCOMES:
Use of prescription medication in the patient's Electronic Health Record at 12 weeks post baseline | EHR data pull at 12 weeks post baseline
  We will look at the patient's medical record from the EHR datapull to cross-reference the self-reported prescription medication use
Use of non-prescription medication in the patient's Electronic Health Record at 12 weeks post baseline | EHR data pull at 12 weeks post baseline
  We will look at the patient's medical record from the EHR datapull to cross-reference the self-reported non-prescription medication use
Results of physical examinations in the patient's Electronic Health Record at 12 weeks post baseline | EHR data pull at 12 weeks post baseline
  We will look at the patient's medical record from the EHR datapull to cross-reference the self-reported pain on average over 7 days at baseline, 8 weeks post baseline, and at 12 weeks post baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Osher Center for Integrative Medicine, Chicago, Illinois, United States